CLINICAL TRIAL: NCT06059248
Title: Effect of Different Head Positions During General Anesthesia Endotracheal Intubation on Postoperative Sore Throat
Brief Title: Effect of Different Head Positions During Endotracheal Intubation on Postoperative Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20230330-05
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Endotracheal Intubation; General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- head sniffing position group (No Intervention): The sniffing position group used the conventional method of endotracheal intubation, the operation method was the same as that of the elevation position group, after the anterior part of the tracheal tube was inserted into the glottis, the head was still kept in the backward position, and the tube core was pulled out by another anesthesiologist (the core extubation force was less than 10N), and the endotracheal tube was inserted at the same time.
- head elevation position group (Experimental): The operation methods of the research group are: left hand laryngoscope, inserted into the laryngeal cavity, fully exposed glottis, right hand tracheal tube from the right corner of the mouth into the mouth, direct vision to insert the anterior part of the endotracheal tube into the glottis, and then the assistant pulls out the tube core (the strength of the extubation core is less than 10N), so that the patient's jaw is adducted, the head remains in the "elevation" position, and the endotracheal tube is inserted at the same time
  Interventions: Other: the head in the "sniffing position "

INTERVENTIONS:
Other: the head in the "sniffing position " — Intubation was performed with the head in the " elevation " position
  Arms: head elevation position group

SUMMARY:
The goal of this [ randomized clinical trial] is to [effect of different head positions on the incidence of postoperative sore throat ] in [patients with endotracheal intubation ]. The main question it aims to answer is: the rate of postoperative sore throat will be reduced or not with the patients' head position changed during intubation.

DETAILED DESCRIPTION:
Objective: To investigate the effect of tracheal intubation in different head positions on the incidence of pharyngeal pain 1, 6 and 24h after operation;Effect of tracheal intubation in different head positions on the incidence of hoarseness 1, 6 and 24h after operation

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing endotracheal intubation abdominal or lower extremity surgery under general anesthesia
2. age 18~65 years old,
3. ASA grade I or II

Exclusion Criteria:

1. patients with pre-existing sore throat or hoarseness before anesthesia;
2. patients with cervical spine disease;
3. patients with upper respiratory infection or a history of tracheostomy;
4. Mallampati score ≥ 3;
5. participation in other clinical trials within the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Rate of Participants with postoperative sore throat | 1, 6, 24 hours after tracheal catheter removal
  Postoperative sore throat is defined as: persistent sore throat with the following grades: 1 point: no sore throat; 2 points: mild, accompanied by odynophagia; 3 points: moderate pain, persistent, worsening with swallowing; 4 points: severe, pain interferes with eating, requires the use of pain medication

SECONDARY OUTCOMES:
Rate of Participants with postoperative hoarseness | 1, 6, 24 hours after tracheal catheter removal
  Hoarseness is defined as a sound quality different from the preoperative voice and is graded as follows: 1 point: none, no hoarseness; 2 points: slight hoarseness, noticed by the patient; 3 points: moderate hoarseness, pronounced to observer; 4 points: severe hoarseness, loss of voice.

CONTACTS AND LOCATIONS:
Overall Officials: Gu Jianping, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kusunoki T, Sawai T, Komasawa N, Shimoyama Y, Minami T. Correlation between extraction force during tracheal intubation stylet removal and postoperative sore throat. J Clin Anesth. 2016 Sep;33:37-40. doi: 10.1016/j.jclinane.2015.12.024. Epub 2016 Apr 6. PMID 27555130
- [Result] Park JJ, Huh H, Yoon SZ, Lim HJ, Go DY, Cho JE, Lee J, Park J, Kim HC. Two-handed jaw thrust decreases postoperative sore throat in patients undergoing double-lumen endobronchial intubation: A randomised study. Eur J Anaesthesiol. 2020 Feb;37(2):105-112. doi: 10.1097/EJA.0000000000001149. PMID 31860598
- [Result] Seo JH, Cho CW, Hong DM, Jeon Y, Bahk JH. The effects of thermal softening of double-lumen endobronchial tubes on postoperative sore throat, hoarseness and vocal cord injuries: a prospective double-blind randomized trial. Br J Anaesth. 2016 Feb;116(2):282-8. doi: 10.1093/bja/aev414. PMID 26787799